CLINICAL TRIAL: NCT05436938
Title: To Evaluate the Mechanism of Jing Si Herbal Tea Liquid Packets and Traditional Western Medicine for Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Sung-Jen Hung, Dermatology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCMF-JCT 111-08
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: DLQI; PHQ-9; PSAI; Serum Cytokine Survey
Keywords: Psoriasis; Psoriatic arthritis; Comorbidities; Jing-Si-Herbal-Tea; Chinese medicine
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Psoriasis patients with mild severity, treatment group (Experimental): with Jing Si herbal tea liquid packets use
  Interventions: Combination Product: Jing Si herbal tea liquid packets use
- Psoriasis patients with mild severity, placebo group (Placebo Comparator): without Jing Si herbal tea liquid packets use
  Interventions: Combination Product: Jing Si herbal tea liquid packets use
- Psoriasis patients with moderate to severe severity, treatment goup (Experimental): with Jing Si herbal tea liquid packets use
  Interventions: Combination Product: Jing Si herbal tea liquid packets use
- Psoriasis patients with moderate to severe severity, placebo group (Placebo Comparator): without Jing Si herbal tea liquid packets use
  Interventions: Combination Product: Jing Si herbal tea liquid packets use

INTERVENTIONS:
Combination Product: Jing Si herbal tea liquid packets use — with or without Jing Si herbal tea liquid packets use

SUMMARY:
Psoriasis is a chronic cutaneous inflammatory disease due to immune dysregulation. It caused skin lesions with thickening plaques and heavy silver scales over the patient's body surface area, including nail deformity, often accompanied by severe itching and pain. Psoriasis is not a contagious or infectious skin disorder, but patients' quality of life is often severely affected by skin symptoms. The annual prevalence of psoriasis in Taiwan is about 0.235%, and about one in 500 people may get psoriasis. Psoriasis has not just skin problems, but it often combines with other comorbidities such as psoriatic arthritis, metabolic syndrome such as diabetes, hypertension, hyperlipidemia and obesity, cardiovascular diseases such as stroke or ischemic heart disease, liver and kidney diseases, inflammatory bowel disease, iritis, and mental illness related to emotional stress and depression. Therefore, patients with psoriasis should regularly receive appropriate therapies to prevent complications and comorbidities. The current standard treatments for psoriasis include traditional topical and systemic treatments, phototherapy, and biologics. Traditional Chinese herbal medicine is also an alternative treatment for psoriasis due to considerable benefits and lower toxicity. Chinese medicine still plays a vital role in the treatment of psoriasis in Taiwanese societies. This experiment will further explore the anti-inflammatory effect of Jing-Si-Herbal-Tea combined with traditional western medicine for three months to reduce inflammatory mediators in the skin and blood and improve the disease severity and quality of life for psoriatic patients.

key words：Psoriasis, Psoriatic arthritis, Comorbidities, Treatment, Jing-Si-Herbal-Tea, Chinese medicine

ELIGIBILITY:
Inclusion Criteria:

- • Subjects were able to give informed consent prior to commencing any trial-related assessments or procedures.

* Subjects were at least 20 years old when they signed the informed consent form.
* At the time of inclusion in this trial, subjects had to have a diagnosis of chronic psoriasis by a dermatologist.
* According to Taiwan's regulations and payment policies, subjects will or have received treatment related to psoriasis. Before being included in the trial, physicians will independently determine the course of treatment with western medicine related to psoriasis.
* The subjects can communicate well with the trial host and understand the contents of the trial case, and follow the trial specifications.
* At the start of the trial, subjects were willing to provide a three-month trial follow-up to record psoriasis severity and dermatological quality of life questionnaires.

Exclusion Criteria:

* The subject is unwilling or unable to comply with the requirements of the trial.
* Subject participated in an interventional clinical trial at this time or within the past 30 days. However, participation in another PMOS (post-marketing observational trial) or registration trial is acceptable.
* Those who are judged by physicians to be infirm, allergic, cold, chronic disease, poor renal function, children under the age of three, children, pregnant, breastfeeding, menstrual period are not suitable to participate in this research.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | 3 months

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | 3 months
Patient Health Questionnaire (PHQ)-9 | 3 months
serum cytokine profiles | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided